## Official Title of the study: Effects of Intermittent Fasting in Metabolic Dysfunction Associated Fatty Liver Disease

NCT number: NCT06664684

Date of the document: 06.05.2022

## Statistical Analysis Plan

Study data were analyzed using SPSS 28.0 software suit. Statistical significance was set at p < 0.05 for all analyses. Data were checked for normality of distribution using the Kolmogorov–Smirnov test. Categorical variables were analyzed using the chi-square test. Median (Quartile 1–Quartile 3) values were used in descriptive statistics. The Mann–Whitney U test was used to determine whether the baseline values were similar between the two groups before the intervention. The before/after comparison of the quantitative data was performed using the Wilcoxon test.